CLINICAL TRIAL: NCT02961855
Title: Double-blinded Multicenter Randomized Clinical Trial to Evaluate the Efficacy and Safety of CLIFE1 and CLIFE2 Gels in Benign Anorectal Surgery
Brief Title: Efficacy and Safety of CLIFE1 Gel in Benign Anorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Viladecans (Other)
Responsible Party: Principal Investigator, María José Linares Gil, Doctor, Hospital de Viladecans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIFE-01FV
Record Dates: First submitted 2016-09-27; First posted 2016-11-11 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Fissure;Anal; Fistula;Rectal; Hemorrhoids
MeSH Terms: conditions — Fissure in Ano; Rectal Fistula; Hemorrhoids | interventions — Anti-Inflammatory Agents; Lidocaine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clife1 gel (lidocaine plus diclofenac) (Experimental): Clife1 gel (lidocaine plus diclofenac) Topical gel containing lidocaine (2%) plus diclofenac (0.5%) (15 g in total) Application of the gel bid from first day post-surgery to day 3 and once daily from day 4 to day 6
  Interventions: Drug: anesthesics plus antiinflammatory, CLIFE1
- Clife2 gel (lidocaine) (Active Comparator): Clife2 gel (lidocaine) Topical gel containing lidocaine (2%) (15 g in total) Application of the gel bid from first day post-surgery to day 3 and once daily from day 4 to day 6
  Interventions: Drug: local anesthesics, CLIFE2

INTERVENTIONS:
Drug: anesthesics plus antiinflammatory, CLIFE1 — anesthesics plus antiinflammatory, CLIFE1 topical gel containing lidocaine plus diclofenac anesthesics plus antiinflammatory
  Other Names: lidocaine plus diclofenac; CLIFE1 topical gel
  Arms: Clife1 gel (lidocaine plus diclofenac)
Drug: local anesthesics, CLIFE2 — local anesthesics, CLIFE2 topical gel containing lidocaine local anesthesics
  Other Names: lidocaine; CLEFE2 topical gel
  Arms: Clife2 gel (lidocaine)

SUMMARY:
Double-blinded multicenter randomized clinical trial to evaluate the efficacy and safety of CLIFE2 (lidocaine, referred as treatment A) respect CLIFE1 (lidocaine plus diclofenac, referred as treatment B) in benign anorectal surgery.

DETAILED DESCRIPTION:
120 patients were randomly assigned to two groups (60 in each group). The study was conducted in two parallel groups, with 1:1 randomization stratified by type of surgery and centre.

Treatment with CLIFE 1 and CLIFE 2 was applied from day 1 to day 6 post-surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing benign anorectal surgery (out or inpatients), with the following diagnoses: anal fissure, fistula, hemorrhoids
* Use of subarachnoid anesthesia with lidocaine

Exclusion Criteria:

* Allergy or Hypersensitivity to lidocaine or other local anesthesics.
* Patients not accepting subarachnoid anesthesia
* Patients with general anesthesia
* Hypersensitivity or contraindication to acetylsalicylic acid.
* History of gastrointestinal hemorrhage or perforation due to nonsteroidal anti-inflammatory drugs (NSAIDs) use
* Active or relapsing peptic ulcer/gastrointestinal hemorrhage
* Serious heart failure.
* Active Crohn disease
* Active ulcerative colitis
* Moderate or sever renal failure
* Severe liver disfunction
* Coagulation disorders requiring treatment with anticoagulant drugs
* Proctitis (due to autoimmune disease, foreign substances, sucally transmitted diseases
* Treatment with: Beta blockers, calcium channel blockers (verapamil and diltiazem), anti-arrhythmics (digoxin, amiodarone), ivabradine, lithium, steroids
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
mean level of pain, as assessed by visual analog scale (VAS) | 3 days post-surgery

SECONDARY OUTCOMES:
Mean level of pain (VAS) at day 3 post-surgery | 6 days post-surgery
Level of pain (VAS), assessed by Andersen scale | 6 days post-surgery
Pain relief | 6 days post-surgery
  Question about pain relief in comparison with the last application (scores from 0 to 4).
analgesics use | 6 days post-surgery
patient satisfaction | 6 days post-surgery
  Satisfaction questionnaire about the efficacy of treatment (6 levels)
demographic and clinical characteristics-1 | baseline
  sex
demographic and clinical characteristics-2 | baseline
  age
safety evaluation as assessed by recording fo adverse events | 6 days post-surgery
  recording of adverse events

IPD SHARING:
Plan to Share IPD: No